CLINICAL TRIAL: NCT03342729
Title: Evaluation of Aging Mastery Program® in Senior Centers Throughout Los Angeles County
Brief Title: Aging Mastery Program® (AMP) Evaluation
Acronym: AMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: The National Council on Aging (Unknown); City of Los Angeles Department of Aging (Unknown); Los Angeles County Area Agency on Aging (Unknown)
Responsible Party: Principal Investigator, Catherine A. Sarkisian, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB #17-000137
Record Dates: First submitted 2017-10-12; First posted 2017-11-17 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Aging; Older Adults; Healthy
MeSH Terms: interventions — Methods

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Immediate exposure to the 10-week Aging Mastery Program (AMP)
  Interventions: Behavioral: Intervention
- Wait-list Group (Placebo Comparator): Class to start 3 months after the Intervention Group
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Intervention — Participants receive the AMP 10-week program immediately
  Arms: Intervention Group
Behavioral: Control — Participants will not received the AMP 10-week program immediately, rather will wait 3-months
  Other Names: Waitlist Control
  Arms: Wait-list Group

SUMMARY:
The Aging Mastery Program® (AMP) is designed to inform, encourage, and support older adults as they take steps to improve their lives and stay engaged in their communities. The program incorporates evidence-informed materials, expert speakers, group discussion, peer support, and small rewards to give participants the skills and tools they need to achieve measurable improvements in managing their health, remaining economically secure, and contributing actively to society. L.A. CAPRA in partnership with the National Council on Aging, City of Los Angeles and the Los Angeles County Department of Aging will evaluate the effectiveness of the AMP program across 5 community-based senior sites. The overall objective of the proposed study is to evaluate the effectiveness of AMP program on improving the health and well-being of older adults using a randomized wait-list controlled trial.

DETAILED DESCRIPTION:
The Aging Mastery Program® (AMP) offers community-based organizations a clear path to engage older adults and address the physical, financial, and emotional wellness of older adults. First piloted nationally in five senior centers, AMP incorporates evidence-based materials, expert speakers, group discussion, and peer support to give participants the skills and tools they need to achieve measurable improvements in managing their health and remaining economically secure. The program aims to empower seniors to make and maintain small, impactful changes to their behaviors to live a healthier, happier, and more secure life. AMP has been field-tested in various rural and urban setting, senior centers, and across an ethnically diverse middle-aged and older adult population, reaching almost 6,000 since 2013. Currently, the program is being evaluated through a quasi-experimental study in New York State and under consideration as an evidence-based program.

The National Council on Aging study team will train six program leads from the City of Los Angeles Department of Aging and Los Angeles Area on Aging to implement Aging Mastery Program® (AMP). The intervention will consist of a 10-week series held once-a-week for an hour and half (90 minutes). It will be group-based and led by trained facilitators and designated expert speakers in a community-based setting (senior centers). The program reviews 10 central areas of aging (1) navigating longer lives, (2) physical activity, (3) sleep, (4) healthy eating and hydration, (5) financial security, (6) medication management, (7) advance care planning, (8) healthy relationships, (9) falls prevention, and (10) community engagement. The intervention is based in social cognitive theory and attribution retraining and incorporates elements such as verbal persuasion, goal setting, problem solving, and attribution retraining techniques that encourage students to adopt controllable and unstable explanations.

Study Participants (N=200 or n=40/site) will be recruited from 5 study sites to participate in the Aging Mastery Program. UCLA study personnel will be on-site to consent older adults to participate in the evaluation of intervention and take part of baseline and post-intervention assessments. Upon signing the consent, study staff will collect self-administered baseline data (measures and measurement tools --i.e. Patient Information Survey, PROMIS and Patient Activation Survey (PAM) from all participants (n=200). After baseline data has been collected, participants will be randomized and assigned to either the immediate intervention groups (n=100 intervention) or the wait-list control (n=100). At each site, forty participants will be in the intervention group and 40 will be in wait-list control. Following the 10-week Aging Mastery Program®, post-intervention assessment (measures and measurement tools --i.e. Patient Information Survey, Patient Satisfaction, PROMIS and PAM) will be administered. During the data collection sessions, study staff will go to community sites and collect post-treatment self-reported assessment

ELIGIBILITY:
Inclusion Criteria:

1. Available to attend the baseline and post-treatment data collection session and subsequent weekly intervention sessions
2. Available to speak and understand English
3. Plans to be living in the region during the next 6 months
4. Has cognitive ability to provide informed consent to participate

Exclusion Criteria:

1. Cannot Speak or Communicate well in English
2. Unavailable to attend the baseline data collection session and subsequent weekly intervention sessions
3. Plans to move away from the region during the next 6 months
4. Lacks cognitive ability to provide informed consent to participate

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-03-15 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
Improvements in health and well-being | Pre-intervention (baseline) and questions will be repeated again 10-weeks after the baseline (for waitlist control/for those in class immediately after the class) as a Post-intervention.
  Patient self-reported questionnaire PROMIS scale; SF-16
Improvements in Patient Activation | Pre-intervention (baseline) and questions will be repeated again 10-weeks after the baseline (for waitlist control/for those in class immediately after the class) as a Post-intervention.
  Patient self-reported questionnaire PAM scale

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Antelope Valley Senior Center, Lancaster, California
  - Freda Mohr Multipurpose Center, Los Angeles, California
  - Potrero Heights Community Center, Montebello, California
  - San Pedro Service Center, San Pedro, California
  - Sherman Oaks East Valley Adult Center, Sherman Oaks, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guerrero LR, Menkin JA, Carrillo CA, Reyes CE, Trejo L, Banks C, Sarkisian CA. Community-Partnered Evaluation of the Aging Mastery Program in Los Angeles Area Senior Centers. Health Educ Behav. 2020 Feb;47(1):57-66. doi: 10.1177/1090198119882992. Epub 2019 Oct 19. PMID 31630566